CLINICAL TRIAL: NCT03329989
Title: A Phase 2 Open-Label Study of EN3835 In The Treatment of Edematous Fibrosclerotic Panniculopathy
Brief Title: Safety and Effectiveness of EN3835 in the Treatment of EFP in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3835-205
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Results first posted 2020-11-23 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-10

CONDITIONS: Edematous Fibrosclerotic Panniculopathy; Cellulite
MeSH Terms: conditions — Cellulite | interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EN3835 Active (Experimental): EN3835 0.84mg (Collagenase Clostridium Histolyticum)
  Interventions: Biological: Collagenase Clostridium Histolyticum

INTERVENTIONS:
Biological: Collagenase Clostridium Histolyticum — During 3 treatment visits 12 injections will be given per treatment area
  Other Names: Xiaflex

SUMMARY:
An open-label study of safety and effectiveness of EN3835 in the treatment of cellulite in adult women.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign and date an informed consent agreement
2. Be a female ≥18 years of age
3. At Screening visit, have at least 2 bilateral quadrants with each quadrant having:

   1. a score of 2 (mild) or greater as reported by the Investigator (CR-PCSS), and
   2. a Hexsel CSS score no greater than 13
4. At Day 1 visit, have assigned bilateral quadrants with each quadrant having:

   1. a score of 2 (mild) or greater as reported by the Investigator (CR-PCSS), and
   2. a Hexsel CSS score no greater than 13
5. Be willing to apply sunscreen to the assigned treatment quadrants before each exposure to the sun while participating in the study (i.e., Screening through end of study)
6. Be judged to be in good health, based upon the results of a medical history, physical examination, and laboratory profile at Screening
7. Have a negative serum pregnancy test at Screening and a negative urine pregnancy test before injection of study drug and be using a stable and effective contraception method (e.g., abstinence, intrauterine device [IUD], hormonal [estrogen/progestin] contraceptives, or double barrier method) for at least 1 menstrual cycle prior to study enrollment and for the duration of the study; or be menopausal defined as 12 months of amenorrhea in the absence of other biological or physiological causes, as determined by the Investigator; or post-menopausal for at least 1 year; or be surgically sterile
8. Be willing and able to cooperate with the requirements of the study
9. Be able to read, complete and understand the patient-reported outcomes rating instruments in English

Exclusion Criteria:

1. Has any of the following systemic conditions:

   1. Coagulation disorder
   2. Evidence or history of malignancy (other than excised basal-cell carcinoma) unless there has been no recurrence in at least 5 years
   3. History of keloidal scarring or abnormal wound healing
   4. Concurrent diseases or conditions that might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the subject's well-being. Any questions about concurrent diseases should be discussed with the Medical Monitor.
   5. Evidence of clinically significant abnormalities on physical examination, vital signs, electrocardiogram (ECG), or clinical laboratory values.
2. Has any of the following local conditions in the area to be treated:

   1. History of lower extremity thrombosis or post-thrombosis syndrome
   2. Vascular disorder (e.g., varicose veins, telangiectasia) in area to be treated
   3. Inflammation or active infection
   4. Active cutaneous alteration including rash, eczema, psoriasis, or skin cancer
   5. Has a tattoo and/or a mole located within 2 cm of the site of injection
3. Requires the following concomitant medications before or during participation in the trial:

   a. Anticoagulant or antiplatelet medication or has received anticoagulant or antiplatelet medication (except for ≤150 mg aspirin daily) within 7 days before injection of study drug
4. Has used any of the following for the treatment of EFP on the legs or buttock within the timelines identified below or intends to use any of the following at any time during the course of the study:

   1. Liposuction in the areas of the body selected for treatment during the 12-month period before injection of study drug
   2. Injections (eg, mesotherapy); radiofrequency device treatments; laser treatment; buttock and/or thigh implant treatment, or surgery (including subcision and/or powered subcision) within the assigned treatment quadrants during the 12-month period before injection of study drug
   3. Endermologie or similar treatments within the assigned treatment quadrants during the 6 month period before injection of study drug
   4. Massage therapy within the assigned treatment quadrants during the 3-month period before injection of study drug
   5. Creams (eg, Celluvera™, TriLastin®) to prevent or mitigate EFP within the assigned treatment quadrants during the 2-week period before injection of study drug
5. Is presently nursing or providing breast milk
6. Intends to become pregnant during the study
7. Intends to initiate an intensive sport or exercise program during the study
8. Intends to initiate a weight reduction program during the study
9. Intends to use tanning spray or tanning booths during the study
10. Has received an investigational drug or treatment within 30 days before injection of study drug
11. Has a known systemic allergy to collagenase or any other excipient of study drug
12. Has received any collagenase treatments at any time prior to treatment
13. Was a subject in a previous cellulite clinical trial of collagenase clostridium histolyticum (CCH) : AUX-CC-830, AUX-CC-831, EN3835-102, EN3835-104, EN3835-201, and/or EN3835-202
14. Any other condition(s) that, in the Investigator's opinion, might indicate the subject to be unsuitable for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female birth gender
Enrollment: 158 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike McLane, PhD, Study Director — Endo Pharmaceuticals
Locations (11):
- United States (11):
  - Endo Clinical Trial Site #1, Scottsdale, Arizona
  - Endo Clinical Trial Site #2, Huntington Beach, California
  - Endo Clinical Trial Site #3, San Diego, California
  - Endo Clinical Trial Site #4, Santa Monica, California
  - Endo Clinical Trial Site #5, Coral Gables, Florida
  - Endo Clinical Trial Site #6, Tampa, Florida
  - Endo Clinical Trial Site #7, West Palm Beach, Florida
  - Endo Clinical Trial Site #8, Alpharetta, Georgia
  - Endo Clinical Trial Site #9, New York, New York
  - Endo Clinical Trial Site #10, Franklin, Tennessee
  - Endo Clinical Trial Site #11, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Collagenase Clostridium Histolyticum (CCH): 12 injections of CCH (Collagenase Clostridium Histolyticum) were administered per treatment area at each treatment visit during 3 visits.
Period: Overall Study
Arm/Group | Collagenase Clostridium Histolyticum (CCH)
Started | 158
Completed | 135
Not Completed | 23
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 8
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Collagenase Clostridium Histolyticum (CCH)
Number analyzed (Participants) | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44
  Not Hispanic or Latino | 114
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 135
  More than one race | 4
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.74 (5.259)
Skin Category (Fitzpatrick Scale) [Count of Participants; unit: Participants]
  I (Pale White) | 3
  II (Fair) | 34
  III (Darker White) | 53
  IV (Light Brown) | 48
  V (Brown) | 10
  VI (Dark Brown) | 10

OUTCOME MEASURES:

1. Primary Outcome: Investigator Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) 2-level Responders
Description: Percentage of responders defined as participants with an improvement in cellulite severity from baseline of at least 2-levels of severity of at least one buttock (left or right) on the Investigator-rated Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) with ratings ranging from "0" (None) to "4" (Severe). A 2-level responder is a participant with a reduction in severity of at least 2-levels from Baseline at that particular visit. Number of participants analyzed is determined by observed participants at each visit.
Time Frame: Day 22, 43, 90, and 180
Population: Effectiveness Population
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH)
Number analyzed (Participants) | 144
Participants
  At Least One of two areas (Left & Right): Day 22: number analyzed (Participants) | 137
  At Least One of two areas (Left & Right): Day 22: Yes | 6
  At Least One of two areas (Left & Right): Day 22: No | 131
  At Least One of two areas (Left & Right): Day 43: number analyzed (Participants) | 133
  At Least One of two areas (Left & Right): Day 43: Yes | 8
  At Least One of two areas (Left & Right): Day 43: No | 125
  At Least One of two areas (Left & Right): Day 90: number analyzed (Participants) | 127
  At Least One of two areas (Left & Right): Day 90: Yes | 17
  At Least One of two areas (Left & Right): Day 90: No | 110
  At Least One of two areas (Left & Right): Day 180: number analyzed (Participants) | 131
  At Least One of two areas (Left & Right): Day 180: Yes | 20
  At Least One of two areas (Left & Right): Day 180: No | 111

2. Secondary Outcome: Investigator Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) 1-level Responders
Description: Percentage of responders defined as participants with an improvement in cellulite severity from baseline of at least 1-level of severity of at least one buttock (left or right) on the Investigator-rated Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) with ratings ranging from "0" (None) to "4" (Severe). A 1-level responder is a participant with a reduction in severity of at least 1-level from Baseline at that particular visit. Percentages are based on the observed counts. Number of participants analyzed is determined by observed participants at each visit.
Time Frame: Day 22, 43, 90, and 180
Population: Effectiveness Population
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH)
Number analyzed (Participants) | 144
Participants
  At Least One of Two Areas (Left & Right): Day 22: number analyzed (Participants) | 137
  At Least One of Two Areas (Left & Right): Day 22: Yes | 55
  At Least One of Two Areas (Left & Right): Day 22: No | 82
  At Least One of Two Areas (Left & Right): Day 43: number analyzed (Participants) | 133
  At Least One of Two Areas (Left & Right): Day 43: Yes | 87
  At Least One of Two Areas (Left & Right): Day 43: No | 46
  At Least One of Two Areas (Left & Right): Day 90: number analyzed (Participants) | 127
  At Least One of Two Areas (Left & Right): Day 90: Yes | 96
  At Least One of Two Areas (Left & Right): Day 90: No | 31
  At Least One of Two Areas (Left & Right): Day 180: number analyzed (Participants) | 131
  At Least One of Two Areas (Left & Right): Day 180: Yes | 90
  At Least One of Two Areas (Left & Right): Day 180: No | 41

3. Secondary Outcome: Subject Satisfaction With Cellulite Treatment Assessment at End of Study
Description: At Day 180, participants rated their satisfaction with cellulite treatment using the 5-point subject satisfaction scale. Ratings range from Very Satisfied with Treatment (2), Satisfied with Treatment (1), Neither Dissatisfied nor Satisfied with Treatment (0), Dissatisfied with Treatment (-1), and Very Dissatisfied with Treatment (-2). Percentages are based on the observed counts.
Time Frame: Day 180
Population: Overall number of participants analyzed is the number participants in effectiveness population at Day 180.
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH)
Number analyzed (Participants) | 130
Participants
  Very Satisfied with Treatment (2) | 25
  Satisfied with Treatment (1) | 48
  Neither Dissatisfied nor Satisfied with Treatment | 32
  Dissatisfied with Treatment (-1) | 12
  Very Dissatisfied with Treatment (-2) | 13

4. Other Pre Specified Outcome: Overall Anti-AUX-I Serum Antibody by Visit
Description: Percent of participants that are seropositive. Descriptive statistics were based on log10 transformation of titer levels. Percentages were based on the number of subjects who had immunogenicity lab samples drawn at the visit. Overall number of participants analyzed is determined by the number of participants in the study. At each visit, the number of participants analyzed is determined by observed participants that had a seropositive sample.
Time Frame: Day 1 to Day 180
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH)
Number analyzed (Participants) | 158
Participants
  Anti-AUX-I: Day 1: number analyzed (Participants) | 156
  Anti-AUX-I: Day 1: Seropositive | 4
  Anti-AUX-I: Day 1: Seronegative | 152
  Anti-AUX-I: Day 22: number analyzed (Participants) | 147
  Anti-AUX-I: Day 22: Seropositive | 104
  Anti-AUX-I: Day 22: Seronegative | 43
  Anti-AUX-I: Day 43: number analyzed (Participants) | 143
  Anti-AUX-I: Day 43: Seropositive | 141
  Anti-AUX-I: Day 43: Seronegative | 2
  Anti-AUX-I: Day 90: number analyzed (Participants) | 134
  Anti-AUX-I: Day 90: Seropositive | 134
  Anti-AUX-I: Day 90: Seronegative | 0
  Anti-AUX-I: Day 180: number analyzed (Participants) | 135
  Anti-AUX-I: Day 180: Seropositive | 134
  Anti-AUX-I: Day 180: Seronegative | 1

5. Other Pre Specified Outcome: Overall Anti-AUX-I Antibody Log Titer Levels by Visit
Description: Descriptive statistics were based on log10 transformation of titer levels. Overall number of participants analyzed is determined by the number of participants in the study. At each visit, the number of participants analyzed is determined by observed participants that had a seropositive sample.
Time Frame: Day 1 to Day 180
Population: Safety Population
Measure: Mean (Standard Deviation); unit: log 10 titer
Arm/Group | Collagenase Clostridium Histolyticum (CCH)
Number analyzed (Participants) | 158
log 10 titer
  Anti-AUX-I: Day 1 positive: number analyzed (Participants) | 4
  Anti-AUX-I: Day 1 positive | 2.046 (1.012)
  Anti-AUX-I: Day 22 positive: number analyzed (Participants) | 104
  Anti-AUX-I: Day 22 positive | 2.268 (1.076)
  Anti-AUX-I: Day 43 positive: number analyzed (Participants) | 141
  Anti-AUX-I: Day 43 positive | 4.681 (0.924)
  Anti-AUX-I: Day 90 positive: number analyzed (Participants) | 134
  Anti-AUX-I: Day 90 positive | 5.937 (0.686)
  Anti-AUX-I: Day 180 positive: number analyzed (Participants) | 134
  Anti-AUX-I: Day 180 positive | 5.556 (0.981)

6. Other Pre Specified Outcome: Overall Anti-AUX-II Serum Antibody by Visit
Description: as for outcome 4
Time Frame: Day 1 to Day 180
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH)
Number analyzed (Participants) | 158
Participants
  Anti-AUX-I: Day 1: number analyzed (Participants) | 156
  Anti-AUX-I: Day 1: Seropositive | 6
  Anti-AUX-I: Day 1: Seronegative | 150
  Anti-AUX-I: Day 22: number analyzed (Participants) | 148
  Anti-AUX-I: Day 22: Seropositive | 50
  Anti-AUX-I: Day 22: Seronegative | 98
  Anti-AUX-I: Day 43: number analyzed (Participants) | 143
  Anti-AUX-I: Day 43: Seropositive | 138
  Anti-AUX-I: Day 43: Seronegative | 5
  Anti-AUX-I: Day 90: number analyzed (Participants) | 131
  Anti-AUX-I: Day 90: Seropositive | 131
  Anti-AUX-I: Day 90: Seronegative | 0
  Anti-AUX-I: Day 180: number analyzed (Participants) | 135
  Anti-AUX-I: Day 180: Seropositive | 130
  Anti-AUX-I: Day 180: Seronegative | 5

7. Other Pre Specified Outcome: Overall Anti-AUX-II Antibody Log Titer Levels by Visit
Description: as for outcome 5
Time Frame: Day 1 to Day 180
Population: Safety Population
Measure: Mean (Standard Deviation); unit: log 10 titer
Arm/Group | Collagenase Clostridium Histolyticum (CCH)
Number analyzed (Participants) | 158
log 10 titer
  Anti-AUX-II: Day 1 positive: number analyzed (Participants) | 6
  Anti-AUX-II: Day 1 positive | 1.607 (0.947)
  Anti-AUX-II: Day 22 positive: number analyzed (Participants) | 50
  Anti-AUX-II: Day 22 positive | 1.942 (1.068)
  Anti-AUX-II: Day 43 positive: number analyzed (Participants) | 138
  Anti-AUX-II: Day 43 positive | 3.641 (1.068)
  Anti-AUX-II: Day 90 positive: number analyzed (Participants) | 131
  Anti-AUX-II: Day 90 positive | 5.255 (0.809)
  Anti-AUX-II: Day 180 positive: number analyzed (Participants) | 130
  Anti-AUX-II: Day 180 positive | 5.141 (0.913)

8. Other Pre Specified Outcome: Anti-AUX-I Neutralizing Antibodies by Visit
Description: A subset of all CCH Treated participants who had positive binding antibody titer levels were tested for the presence or absence of Neutralizing Antibodies. Overall Number of Participants Analyzed is determined by the number of participants in the highest and lowest quartiles at Day 90 (Q1 and Q4) of seropositive participants at each of two visits (Day 90 and Day 180).
Time Frame: Day 1 to Day 180
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH)
Number analyzed (Participants) | 34
Participants
  anti-AUX-I Neutralizing Antibody: Day 1: number analyzed (Participants) | 1
  anti-AUX-I Neutralizing Antibody: Day 1: Positive | 0
  anti-AUX-I Neutralizing Antibody: Day 1: Negative | 1
  anti-AUX-I Neutralizing Antibody: Day 90: Positive | 26
  anti-AUX-I Neutralizing Antibody: Day 90: Negative | 8
  anti-AUX-I Neutralizing Antibody: Day 180: number analyzed (Participants) | 33
  anti-AUX-I Neutralizing Antibody: Day 180: Positive | 19
  anti-AUX-I Neutralizing Antibody: Day 180: Negative | 14

9. Other Pre Specified Outcome: Anti-AUX-II Neutralizing Antibodies by Visit
Description: A subset of all CCH Treated participants who had positive binding antibody titer levels were tested for the presence or absence of Neutralizing Antibodies. Overall Number of Participants Analyzed is determined by the number of participants in the study. Number of Participants Analyzed is determined by observed participants that had a seropositive sample at each visit and the antibody level at Day 71 in Q1 and Q4.
Time Frame: Day 1 to Day 180
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Clostridium Histolyticum (CCH)
Number analyzed (Participants) | 32
Participants
  anti-AUX-II Neutralizing Antibodies: Day 1: number analyzed (Participants) | 1
  anti-AUX-II Neutralizing Antibodies: Day 1: Positive | 1
  anti-AUX-II Neutralizing Antibodies: Day 1: Negative | 0
  anti-AUX-II Neutralizing Antibodies: Day 90: Positive | 24
  anti-AUX-II Neutralizing Antibodies: Day 90: Negative | 8
  anti-AUX-II Neutralizing Antibodies: Day 180: number analyzed (Participants) | 31
  anti-AUX-II Neutralizing Antibodies: Day 180: Positive | 20
  anti-AUX-II Neutralizing Antibodies: Day 180: Negative | 11

ADVERSE EVENTS:
Time Frame: All (serious and non-serious) AEs, from Day 1 up to Day 180
Description: All (serious and nonserious) AEs, whether elicited or observed during study visits or spontaneously reported by the participant, including events that occurred from the time the participant signed the study-specific consent form until completion of or discharge from the study.
Groups:
- Collagenase Clostridium Histolyticum (CCH): EN3835 0.84mg (Collagenase Clostridium Histolyticum)
  Collagenase Clostridium Histolyticum: During 3 treatment visits 12 injections is given per treatment area
Arm/Group | Collagenase Clostridium Histolyticum (CCH)
All-Cause Mortality (participants affected / at risk) | 0/158
Serious Adverse Events (participants affected / at risk) | 1/158
Other Adverse Events (participants affected / at risk) | 158/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Collagenase Clostridium Histolyticum (CCH) (N=158)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Collagenase Clostridium Histolyticum (CCH) (N=158)
Injection site bruising (General disorders) | 136
Injection site pain (General disorders) | 76
Injection site swelling (General disorders) | 35
Injection site pruritus (General disorders) | 27
Injection site discolouration (General disorders) | 26
Injection site nodule (General disorders) | 23
Injection site warmth (General disorders) | 18
Injection site haemorrhage (General disorders) | 17
Injection site mass (General disorders) | 10
Hemosiderin stain (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/89/NCT03329989/Prot_001.pdf
  • Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT03329989/SAP_002.pdf